CLINICAL TRIAL: NCT07356414
Title: "SwallowFit," an Exercise Program and Randomized Clinical Trial Designed for US Service Members, Veterans, and Families Affected by Parkinson's Disease.
Brief Title: SwallowFIT Study in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Giselle Carnaby, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001444; FY24 HT942524PRPIIRA (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Swallowing; US Service members; Veterans; SwallowFIT
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A single site, double blind randomized controlled trial comparing a proactive swallow exercise intervention to a control group receiving clinical monitoring only (or CMO).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study investigators (PI, Co-I's, and Biostatistician), study coordinator and the Independent Evaluator, will be blind to the treatment allocation of the subjects. The PI will evaluate de-identified videoed assessments, and swallowing videofluoroscopic data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SwallowFit Intervention (Experimental): Subjects randomized to intervention will receive 6-weeks of twice weekly SwallowFIT per protocol (1-hour session each day). The program begins with provision of general education on swallowing and swallowing change from the Parkinson's Foundation and Michael J Fox association websites. Following this the program trains a modified effortful swallow technique at its onset using surface electromyographic (sEMG) biofeedback to guide the development of better swallow movement form, effort and performance. From there it applies a hierarchy of swallowing exercises/tasks involving swallowing food/fluid materials at different complexity levels (swallow specificity) to stimulate and train progressive resistance and leverage variability of coordinated speeded actions.
  Interventions: Behavioral: SwallowFit
- Clinical Monitoring Only (CMO) (No Intervention): CMO intervention reflects current swallow management practice for PD, where physicians monitor clinical function in swallowing and other related symptomology, referring for swallowing treatment only if an obvious issue has been identified. Subjects randomized to CMO will also receive general education on swallowing and swallow changes from the Parkinson's Foundation and Michael J Fox association websites.

INTERVENTIONS:
Behavioral: SwallowFit — The SwallowFIT protocol follows an increasing task difficulty (levels on the hierarchy) and motor learning strategy. Progression on the hierarchy is guided and monitored by the occurrence of inefficiency markers in swallow wing (e.g. excessive lingual pumping, swallow hesitation, throat clearing etc.) confirmed from the baseline clinical and video fluoroscopic evaluations.
  Other Names: Swallowing exercises
  Arms: SwallowFit Intervention

SUMMARY:
The goal of this clinical trial is to learn if a proactive swallow exercise will help to improve swallow fitness in patients with Parkinson's disease.

The aim of the study is to assess how effective this exercise is and to measure the change in swallowing fitness from the beginning to the end of the study.

Patients who are given the exercise training will be compared to participants who are treated using the usual standard treatment.

Patients will have 6 weeks of twice-weekly SwallowFIT training. Each session will be an hour long.

DETAILED DESCRIPTION:
SwallowFIT: Subjects will receive 6-weeks of twice weekly SwallowFIT intervention per protocol (1-hour session each visit) from the BAMC speech language Pathologist (study SLP) at BAMC. Completion of the program will include 12 visits. The program is designed from a previous successful pilot trial. It begins with provision of general education on swallowing and swallowing change from the Parkinson's Foundation and Michael J Fox association websites.

Following this the program trains a modified effortful swallow technique at its onset using sEMG to guide the development of better swallow movement form, effort and performance. Once swallowing form is established, the program uses a hierarchy of swallowing tasks involving swallowing food/fluid materials at different complexity levels (swallow specificity) to stimulate and train progressive resistance and leverage variability of coordinated speeded actions.

Clinical Monitoring Only (CMO): This intervention mirrors the experimental intervention in all aspects, but the treatment type applied. CMO intervention reflects current swallow management practice for PD, where physicians monitor clinical function in swallowing and other related symptomology, referring for swallowing treatment only once an obvious issue has been identified.

ELIGIBILITY:
Inclusion Criteria:

1. Adult S-VWP between >35-90 years of age
2. Diagnosis of Idiopathic Parkinson's Disease [IDP] (either or suspected, tremor-predominant or rigid predominant)
3. Disability level of Hoehn & Yahr stages II-III as indicated in their most recent neurological evaluation
4. Swallowing concern, confirmed by Modified Unified Parkinson Disease Rating Scale [MDS-UPDRS]-
5. ADL swallowing item >0, or Mann Assessment of Swallowing scale [MASA] score ≤185.
6. Able to consume oral nutrition [Functional Oral Intake Score ≤ 6]
7. Ambulatory
8. No change of medication for at least 4 weeks before study inclusion

Exclusion Criteria:

1. Classified as Hoehn and Yahr stages IV
2. Unable to follow 2 step commands
3. History of other neurological disease potentially causing dysphagia
4. Dementia (MMSE<20; Montreal cognitive assessment (MoCA) ≤ 20)
5. Severe depression (BDI>19)
6. Severe dyskinesia of head and neck (resulting in problems with MBSS recording)
7. Severe documented Gastrointestinal disease
8. History of Gastro-esophageal surgery
9. History of Head or neck cancer with swallowing impairment or surgical intervention
10. History of breathing disorders or diseases (e.g., Asthma, chronic obstructive pulmonary disease (COPD) requiring assistive breathing support.
11. Untreated hypertension
12. Heart disease requiring restricted activity and medical intervention
13. Speech therapy intervention for swallowing within the past three months
14. Women who are pregnant, nursing, or who plan to become pregnant during the study

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-06-29 (Estimated)

PRIMARY OUTCOMES:
Mann Assessment of Swallowing Ability (MASA) | Baseline to 6 months
  The MASA score is measured using a 5-point to 10-point rating scale. The total possible score of the MASA is 200 points, and the cutoff value is 177 points. The results of the MASA are interpreted as no abnormality (≥178), mild dysphagia (168-177), moderate dysphagia (139-167), and severe dysphagia (≤138).
Modified Unified Parkinson Disease Rating Scale (MDS-UPDRS) | Baseline to 6 months
  The MDS-UPDRS uses a 0-4 scoring system, with higher scores indicating more severe symptoms. Parts I-III are scored on a 0-4 scale, while Part IV uses "yes" and "no" ratings. The total score range is 0-260, with 0 representing no disability and 260 representing total disability.
Modified Hoehn and Yahr (HY) Scale | Baseline to 6 months
  The Hoehn and Yahr (H&Y) scale is a grading system used to assess the progression and severity of motor symptoms in Parkinson's disease (PD). It ranges from Stage 0 (no signs of disease) to Stage 5 (severe disability, wheelchair or bed bound). Stages 1, 1.5, 2, and 2.5 are considered early stages, while stages 3, 4, and 5 represent later, more advanced stages.
Montreal Cognitive Assessment (MoCA) | Baseline to 6 months
  The Montreal Cognitive Assessment (MoCA) is a cognitive screening tool with a maximum score of 30 points, with a score of 26 or higher generally indicating normal cognitive function. Scores between 18 and 25 may suggest mild cognitive impairment (MCI), while scores below 18 may indicate moderate to severe impairment.
PD Quality of Life Scale (PDQ-39) | Baseline to 6 months
  The PDQ-39 is a questionnaire used to assess the impact of Parkinson's disease on quality of life. It consists of 39 questions, each rated on a 5-point scale from 0 (never) to 4 (always). Scores for the 39 questions are added to obtain a total score.
  The scores for the 8 subscales (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and physical discomfort) are obtained by summing the scores for the relevant questions within each subscale.
  The total score and subscale scores range from 0 to 100, with higher scores indicating a greater impact of Parkinson's disease on quality of life.

SECONDARY OUTCOMES:
Modified Barium Swallowing Impairment Profile, overall impression score (MBSImp OI score) | Baseline to 6 months
  In the context of the Modified Barium Swallow Impairment Profile (MBSImP), Overall Impression (OI) scoring is the most common method used to assess swallowing physiology. It involves assigning a score to each of the 17 physiological components based on the most severe impairment observed across different swallowing tasks. These scores range from 0 to 4 depending on the component, and total scores range from 0-68 with higher scores indicating greater impairment.
Spontaneous Swallowing Frequency (SSF) | Baseline to 6 months
  Spontaneous swallowing frequency (SSF) scoring refers to counting the number of times a person swallows without any specific prompting or external stimuli. It's a method used to assess swallowing function, particularly in conditions like dysphagia (difficulty swallowing), and can be a tool for screening and evaluating swallowing problems. A 5-10 minute sampling window is often used to calculate SSF.
  Healthy Swallowing:
  In healthy individuals, spontaneous swallowing typically occurs at a rate of 1-2 swallows per minute.
  Dysphagia:
  Patients with dysphagia often have a reduced SSF compared to healthy individuals.
  Thresholds:
  Some studies have suggested a threshold of 0.40 swallows per minute as a potential indicator of significant dysphagia.
Penetration Aspiration Scale (PAS) | Baseline to 6 months
  The Penetration-Aspiration Scale (PAS) is an 8-point scale used to assess the depth and response to airway invasion during swallowing. It helps clinicians and researchers understand the severity of swallowing dysfunction by categorizing the location of the bolus within the airway and whether it's expelled or not. The scale is used in videofluoroscopic swallowing studies (VFSS) to quantify swallowing event. A score of 1 would indicate no material entered the airway while a score of 8 would indicate the most amount of material aspirated during swallowing.
Analysis of Swallowing Physiology: Events, Kinematics and Timing (ASPEKT) | Baseline to 6 months
  Method of measuring physiologic kinematics and timing for swallowing images retrieved from modified barium swallow (MBSS). It evaluates of 8 key parameters of swallowing taken by frame analysis on open-source NIH, Image J software. Scoring of kinematic swallow movements will be evaluated using the published protocol
Functional Oral Intake Scale (FOIS) | Baseline to 6 months
  The Functional Oral Intake Scale (FOIS) is a 7-point ordinal scale used to assess a patient's ability to swallow and eat safely and efficiently. Scores range from 1 to 7, with higher scores indicating better swallowing function and a greater ability to participate in oral intake.
Lingual Pressure/movement | Baseline to 6 months
  The Lingual Pressure Movement Scale, part of the AIMS (Abnormal Involuntary Movement Scale), assesses the severity of tongue movements. It uses a 0-4 scale, where 0 represents no movement, 1 represents minimal movement (may be extreme normal), 2 represents mild movement, 3 represents moderate movement, and 4 represents severe movement.
Sydney Swallowing Questionnaire (SSQ) | Baseline to 6 months
  The Sydney Swallow Questionnaire (SSQ) is scored by summing the individual scores for each question. It consists of 17 questions, with most questions scored on a visual analog scale (VAS), ranging from 0 to 100 mm. The total possible score is 1700. Higher scores indicate more severe swallowing difficulties.
Protocol Adherence Measure | Baseline to 6 months
  Percentage attendance measured by number of prescribed exercise sessions completed
Patient Perception of Swallowing (VAS) | Baseline to 6 months
  In patient perception of swallowing, a Visual Analogue Scale (VAS) is used to assess a patient's subjective experience of swallowing difficulties. Patients mark a point on a line (typically 100 mm) that represents the severity of their swallowing problem, with 0 indicating no trouble and 100 indicating a total inability to swallow.
Patient/Caregiver Acceptability/Satisfaction Scale (PA/SS) | Baseline to 6 months
  A 5 item scale where each item is scored on a Likert scale from 0-10. Total scores range from 0-50 with a higher score indicating that the SwallowFIT program was more helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Carnaby, PhD, MP, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Brooke Army Medical Center (BAMC), San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will report and publish in a peer-reviewed journal (trials journal) the study protocol and proposed analysis, to provide similar information to the national and international scientific community.
  Information provision and awareness-raising will take place during project inception and intensify as results become available.
  Study results will be published and displayed on the project webpage following completion of the 6 month follow up of all subjects.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study is complete and unblinded, the study team will submit all remaining scientific data to the data repository, and we will update the study status to "completed" in clinical trials.gov. According to the study timeline, all generated scientific data will approximately coincide with the submission of the results to clinicaltrials.gov and will occur no later than by the end of award. Scientific data included in published manuscripts will be available at the time of publication. According to the proposed project timeline, all generated scientific data will approximately coincide with the submission of the results to clinicaltrials.gov at the end of the award, and full data sharing (via repository) will occur no later than six months after completion of the study or acceptance for publication of the main findings from the final dataset.

REFERENCES:
- See also: Lab website for Principle Investigator regarding the study. — https://labs.uthscsa.edu/saul/